CLINICAL TRIAL: NCT05485597
Title: Usability and Feasibility Study of Myosuit-based Gait Training for Ambulatory Neurological Patients With Gait Disorders
Brief Title: Myosuit-based Gait Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rehaklinik Zihlschlacht AG (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RZS_05_2022
Record Dates: First submitted 2022-07-26; First posted 2022-08-03 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Neurologic Gait Disorder
Keywords: Exosuit; Training; Rehabilitation
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: The proposed trial is designed as an open-label, non-randomized interventional study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group: Neurological inpatients with Gait disorders (Experimental): The group participates in the study intervention (they will undergo the Myosuit-based gait training)
  Interventions: Device: Myosuit-based gait training

INTERVENTIONS:
Device: Myosuit-based gait training — In a period of four weeks participants will undergo eight individual task-specific overground gait training sessions with the Myosuit. The sessions will be started with a therapist, and if possible and as soon as possible, the patient will train with an assistant. During the therapy sessions, the patient will be asked to perform various task-specific exercises with the Myosuit, such as Sit-to-stand-, Balance- and walking exercises. Depending on the individual skill level of the participant, a higher level of difficulty in task-specific exercises can be performed. The training sessions are set to last 45 minutes. All training sessions will be accompanied by a certified (physio)therapist or trained assistant and a study investigator.

SUMMARY:
This study will investigate the safety and feasibility of over-ground training sessions with the Myosuit for the neurological inpatients of rehabilitation clinic Zihlschlacht with a gait disorder and their therapists. It will also examine the acceptability and motivation of patients and therapists to use the device for training in the clinical setting and at home or community level. Moreover, it will present first results of the training efficacy with the Myosuit in the inpatient setting on the mobility level of the International Classification of Function. The proposed trial is designed as an open-label, non-randomized interventional study

DETAILED DESCRIPTION:
Neurological disorders are the leading cause of long-term disability in adults worldwide. The activity most affected by a neurological disease is walking. Gait disorders occur in approximately 60% of patients hospitalized for a neurological disease and are the first step toward immobility and loss of independence. Not reaching the walking speed, which is necessary to walk safely outside, hinders social (re)integration and the ability to participate in society. As a result, many neurological patients with gait disorders experience a significantly reduced health-related quality of life. Soft, lightweight wearable robots appear to be good candidates for supporting physical therapy in a clinical environment and improving functional mobility in outdoor settings and as assistive devices during activities of daily living within a home-based environment. The integration of these robots into home-based rehabilitation programs could greatly contribute to increasing the patient's activity level and social interaction, which increases the health-related quality of life in chronic neurological patients. The Investigators want to integrate this new form of therapy in the rehabilitation programme from inpatient to home setting with the aim of maintaining and/or improving patients' functional ambulatory ability and enable them to perform activities of daily living more independently. This research aims to evaluate the usability of the innovative wearable robot 'the Myosuit" and the feasibility of this new form of therapy in the inpatient setting. The investigators will also measure qualitatively and quantitatively the patients' motivation to want to continue using the device for the home training and the staff's motivation to recommend the training with this device in the home setting. Furthermore, the investigators will evaluate the staff's judgment on the feasibility of recommending the Myosuit for home-training.

In a time period of four weeks participants will undergo eight individual task-specific overground gait training sessions with the Myosuit.The inpatient training sessions will be started with a therapist, and if possible and as soon as possible, the patient will continue training with an assistant of therapy. Both therapists and assistants will be trained with the device before the study begins. The investigators introduce the training with assistants as an important step for transferring the inpatient training to the home setting where the relatives will assist the patients in the training with the Myosuit and they will have no background in physiotherapy as it is the case of the assistants in this study. The investigators assume that if the inpatient training is possible with therapists and subsequently with the assistants, it will be certainly feasible with the relatives.

For this study, the Myosuit (MyoSwiss AG, Zurich, Switzerland) will be used. The Myosuit is CE-Marked (Conformité Européenne; in accordance with European legislation), with reference number 1910001. The Myosuit is an untethered wearable robot designed to assist the essential mobility functions across activities of daily life, such as walking, standing, sitting, making transfers or climbing stairs. The Myosuit actively supports knee and hip extension in the early- to mid-stance phase of the gait cycle and passively aids hip flexion during swing, using elastic rubber bands

All the participants will be recruited from inpatients of Rehabilitation clinic Zihlschlacht by qualified (physio)therapists. The study participants will receive sufficient information about the study design and the risks and benefits of their participation. Patients have to meet defined physical requirements. To screen whether the patients meet these physical (manufacturer's recommendations) requirements, for the safety and feasibility of using the Myosuit, a clinical evaluation will be undertaken prior to the training period. In addition, to be included in the study, participants must meet the study inclusion and exclusion criteria It is planned to recruit 15 ambulatory neurological patients with gait disorder. The estimated duration is 5 months.

Mainly descriptive statistics will be performed in order to analyze the obtained data. Normal distribution will be determined visually by quantile-quantile plots and numerically by Shapiro-Wilk Normality Test. Matched-paired tests will be used to examine differences in pre-test and post-test scores. Associations between paired samples will be measured by either Spearman's rho or Pearson correlation coefficient depending on normality. Effect size will be calculated in order to measure meaningful differences between pre-test and post-test scores. A two-sided p value of <0.05 is considered statistically significant. All analyses are going to be performed using IBM® SPSS® Statistics and MATLAB and Statistics Toolbox, The MathWorks, Inc., Natick, Massachusetts, United States.

ELIGIBILITY:
Inclusion Criteria:

* FAC score between 2 and 4
* Intact or mildly to moderately impaired cognition: Mini Mental State Examination (MMSE) score above 17 points
* Subject is at least 18 years old
* A height between 150 cm and 195 cm
* A weight between 45 to 110 kg

Exclusion Criteria:

* Specific neurological disorders such as Parkinson's disease and Multiple sclerosis
* Neurological patients without gait disorders
* Unstable cardiovascular and respiratory conditions
* Functional Reach Test < 15.24 cm
* 10MWT not possible with the assistance of a person
* Major musculoskeletal conditions (e.g., rheumatoid arthritis), major limited lower extremity's range of motion, orthopedic problems and/or significant lower extremity joint pain that could affect the application of the Myosuit
* Significant lower limb contractures (knee flexion or hip flexion contracture of >10°, Varus deformity >10°, Valgus deformity >10°) that could affect the application of the Myosuit
* Skin integrity (on surfaces that would contact the device)
* Significant osteoporosis (bone fragility) assessed by a medical doctor
* Pregnancy
* Incapacity to (safely) understand and/or follow instructions (e.g., aphasia, limited knowledge of German)
* Incapacity to understand formal consent
* Currently participating in other (internal) interventional studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Usability of the Myosuit during task specific training | 4 weeks
  The usability will be measured with the System Usability Scale (SUS). The SUS questionnaire will be completed by the participants, as well as therapists and therapy assistants. The SUS is an easy, valid and reliable tool for measuring the usability of a device. It consists of a 10-item questionnaire about the usability of a device with five response options for respondents; from strongly agree to strongly disagree. A score above 68 can be considered above average and anything below 68 is below average.
Usability of the Myosuit during task specific training | 4 weeks
  The usability will be measured with the Usefulness, Satisfaction, and Ease of use Questionnaire (USE). The USE questionnaire will be completed by the participants, as well as therapists and therapy assistants. The USE measures the subjective usability of a product or service. It is a 30-item questionnaire that examines four dimensions of usability: usability, ease of use, ease of learning, and satisfaction. a higher score indicates better usability.
Safety of the Myosuit during task specific training. | 4 weeks
  The safety will be analyzed by the risk of falling (near falls, falls and adverse events (AE)) and the change in walking speed, step length and cadence while performing the 10 Meter Walk Test (10MWT) with versus without the Myosuit.

SECONDARY OUTCOMES:
Motivation of patients to use the Myosuit during and after their inpatient rehabilitation | 4 weeks
  The motivation will be measured by conducting an interview with the participants
Motivation of therapists to use the Myosuit as a facilitator for gait training. | 4 weeks
  The motivation will be measured by conducting an interview with the therapists
Motivation of therapy assistants to use the Myosuit as a facilitator for gait training. | 4 weeks
  The motivation will be measured by conducting an interview with the therapy assistants
Efficacy of the four-week Myosuit-based gait training on mobility | 4 weeks
  The mobility will be measured by the de Morton Mobility Index (DEMMI). The DEMMI is an assessment on an ordinal scale level, which can depict the mobility status of geriatric patients across the entire mobility spectrum by means of 15 items. It is hierarchically structured from easy to difficult. In five subcategories (bed, chair, static balance, walking, and dynamic balance) different activities are tested. Most items are rated with zero points or one point, depending on whether the activity can be performed (1) or not (0). For some items, a maximum of two points can be awarded in order to evaluate the level of support or the quantity of walking distance in a more differentiated way. The tester adds up the points to a raw score (max. 19 points) and converts this into the DEMMI score (0 to 100 points) for statistical reasons using a conversion table. In general, a higher score indicates better mobility.
Efficacy of the four-week Myosuit-based gait training on walking speed | 4 weeks
  The walking parameter walking speed will be measured by the 10-Meter Walk Test (10MWT). The 10MWT is a performance measure used to assess walking speed in meters per second over a short distance. Walking speed < 0.70 m/s is indicative of increased risk of adverse events (fall, hospitalisation, fracture, etc.). A speed <0.40 m/s indicates a household ambulator, a speed between 0.40 and 0.80 m/s indicates a limited community ambulator and speed > 0.80 m/s indicates the possibility of a community ambulator.
Efficacy of the four-week Myosuit-based gait training on walking capacity | 4 weeks
  The walking parameter walking capacity will be measured by the 6-Minute Walk Test (6MWT). The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. An increase in the walked distance indicates improvement in basic mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehaklinik Zihlschlacht AG, Zihlschlacht-Sitterdorf, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haufe FL, Kober AM, Schmidt K, Sancho-Puchades A, Duarte JE, Wolf P, Riener R. User-driven walking assistance: first experimental results using the MyoSuit. IEEE Int Conf Rehabil Robot. 2019 Jun;2019:944-949. doi: 10.1109/ICORR.2019.8779375. PMID 31374751
- [Result] Haufe FL, Schmidt K, Duarte JE, Wolf P, Riener R, Xiloyannis M. Activity-based training with the Myosuit: a safety and feasibility study across diverse gait disorders. J Neuroeng Rehabil. 2020 Oct 8;17(1):135. doi: 10.1186/s12984-020-00765-4. PMID 33032627
- [Result] Wright A, Stone K, Martinelli L, Fryer S, Smith G, Lambrick D, Stoner L, Jobson S, Faulkner J. Effect of combined home-based, overground robotic-assisted gait training and usual physiotherapy on clinical functional outcomes in people with chronic stroke: A randomized controlled trial. Clin Rehabil. 2021 Jun;35(6):882-893. doi: 10.1177/0269215520984133. Epub 2020 Dec 27. PMID 33356519
- [Result] Buesing C, Fisch G, O'Donnell M, Shahidi I, Thomas L, Mummidisetty CK, Williams KJ, Takahashi H, Rymer WZ, Jayaraman A. Effects of a wearable exoskeleton stride management assist system (SMA(R)) on spatiotemporal gait characteristics in individuals after stroke: a randomized controlled trial. J Neuroeng Rehabil. 2015 Aug 20;12:69. doi: 10.1186/s12984-015-0062-0. PMID 26289955
- [Result] Mehrholz J, Thomas S, Werner C, Kugler J, Pohl M, Elsner B. Electromechanical-assisted training for walking after stroke. Cochrane Database Syst Rev. 2017 May 10;5(5):CD006185. doi: 10.1002/14651858.CD006185.pub4. PMID 28488268